CLINICAL TRIAL: NCT00887250
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Clinical Study to Evaluate the Antihypertensive Efficacy and Safety of Losartan (MK954, DuP753) in Patients With Mild to
Brief Title: A Study to Investigate the Antihypertensive Efficacy of MK0954
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009_580; MK0954-050
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2009-06-24 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo
- 2 (Experimental): Losartan 50 mg for 12 weeks
  Interventions: Drug: losartan potassium
- 3 (Experimental): Losartan 50 mg titrated to 100 mg after 6 weeks
  Interventions: Drug: Comparator: losartan

INTERVENTIONS:
Drug: losartan potassium — 50 mg Losartan (MK0954) tablet taken once daily for 12 weeks.
  Other Names: MK0954
  Arms: 2
Drug: Comparator: losartan — 50 mg tablet of Losartan (MK0954) taken once daily for 6 weeks, Non-responders will then have the dose up titrated to 100 mg for remaining 6 weeks.
  Other Names: MK0954
  Arms: 3
Drug: Comparator: Placebo — Placebo to Losartan
  Arms: 1

SUMMARY:
After a 4 week placebo period, patients were randomized to Placebo or Losartan 50 mg arms, after 6 weeks non-responders were up titrated to 100 mg losartan for the remaining 6 weeks. This study evaluated if losartan is more effective than placebo in lowering sitting diastolic blood pressure and is well tolerated in patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with mild to moderate hypertension (SDBP 95-115 mm Hg)
* Patient has no medical problems or treatments that might effect their blood pressure

Exclusion Criteria:

* Pregnant or lactating females
* Patient has secondary hypertension or malignant hypertension
* Sitting systolic blood pressure > 210 mm Hg
* History of stroke
* History of myocardial infarction with in past year
* Current or prior history of heart failure
* Known hypersensitivity to losartan
* Prior exposure to losartan
* Patients known to be HIV positive
* Patient is abusing or has abused alcohol or other drugs within the past 4 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 1991-12; Primary Completion 1992-08 (Actual); Study Completion 1992-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 22 sites in the United States. Prime Therapy Period: December, 1991 to August, 1992.
Pre-assignment Details: Patients could be randomized after the 4-week placebo baseline period if their mean sitting diastolic blood pressure (SiDBP) was 95-115 mm Hg and ≤7 mm Hg from the mean SiDBP after 2 weeks of placebo therapy
Groups:
- Placebo: Losartan placebo orally once daily for 12 weeks
- Losartan 50 mg: Losartan 50 mg orally once daily for 12 weeks
- Losartan 50/100 mg: Losartan orally once daily for 12 weeks, initiated as 50 mg and titrated to 100 mg for nonresponders (SiDBP ≥90 mm Hg) after 6 weeks
Period: Overall Study
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Started | 116 | 127 | 123
Completed | 98 | 115 | 110
Not Completed | 18 | 12 | 13
Not completed — Adverse Event | 3 | 0 | 7
Not completed — Lack of Efficacy | 9 | 6 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Patient uncooperative | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg | Total
Number analyzed (Participants) | 116 | 127 | 123 | 366
Age Continuous [Mean (Full Range); unit: years] | 53.8 [26 to 78] | 53.2 [28 to 75] | 55.1 [28 to 76] | 54.0 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 45 | 131
  Male | 74 | 83 | 78 | 235
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 92 | 104 | 101 | 297
  Black | 17 | 14 | 16 | 47
  Hispanic | 7 | 8 | 4 | 19
  Indian | 0 | 1 | 0 | 1
  Oriental | 0 | 0 | 2 | 2
Sitting Diastolic Blood Pressure (SiDBP) [Mean (Full Range); unit: mm Hg] | 101.3 [95 to 115] | 102.2 [95 to 113] | 102.2 [95 to 114] | 101.9 [95 to 114]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Mean change from baseline in trough (24 hours post dose) SiDBP at Week 12
Time Frame: At baseline and at 12 weeks (24 hours post dose)
Population: The primary analysis employed an "all patients treated" approach that included patients with at least one treatment period measurement. The last measurements of withdrawn patients were carried forward to subsequent timepoints. Missing data were estimated by carrying forward data from the last visit (excluding baseline) at which it was available.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Number analyzed (Participants) | 114 | 125 | 118
mm Hg | -4.3 (6.7) | -7.9 (7.6) | -8.6 (7.7)

2. Secondary Outcome: Categories of Hypertensive Response in Trough Diastolic Blood Pressure (SiDBP) at Week 6
Description: Patients with trough SiDBP <90 mm Hg were in Category I, ≥90 but decreased at least 10 mm Hg were in Category II, and ≥90 and decreased less than 10 mm Hg were in Category III.
Time Frame: 24 hours post dose at Week 6
Population: An "all patients treated" approach was employed that included patients with at least one treatment period measurement. The last measurements of withdrawn patients were carried forward to subsequent timepoints. Missing data were estimated by carrying forward data from the last visit (excluding baseline) at which it was available.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Number analyzed (Participants) | 114 | 125 | 118
Participants
  Category I | 14 | 37 | 37
  Category II | 8 | 20 | 21
  Category III | 92 | 68 | 60

3. Secondary Outcome: Categories of Hypertensive Response in Trough Diastolic Blood Pressure (SiDBP) at Week 12
Description: as for outcome 2
Time Frame: 24 hours post dose at Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Number analyzed (Participants) | 114 | 125 | 118
Participants
  Category I | 19 | 40 | 37
  Category II | 12 | 18 | 24
  Category III | 83 | 67 | 57

4. Secondary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 6
Description: Mean change from baseline in trough (24 hours post dose) SiDBP at Week 6
Time Frame: At baseline and at 6 weeks (24 hours post dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Number analyzed (Participants) | 114 | 125 | 118
mm Hg | -3.5 (5.8) | -6.9 (7.0) | -7.9 (7.1)

5. Secondary Outcome: Mean Change From Baseline in Peak Sitting Diastolic Blood Pressure (SiDBP) at Week 6
Description: Mean change from baseline in peak (6 hours post dose) SiDBP at Week 6
Time Frame: At baseline and at 6 weeks (24 hours post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Number analyzed (Participants) | 108 | 118 | 111
mm Hg | -4.1 (6.9) | -9.7 (8.7) | -8.9 (8.7)

6. Secondary Outcome: Mean Change From Baseline in Peak Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Mean change from baseline in peak (6 hours post dose) SiDBP at Week 12
Time Frame: At baseline and at 12 weeks (6 hours post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 50 mg | Losartan 50/100 mg
Number analyzed (Participants) | 108 | 121 | 113
mm Hg | -4.7 (7.9) | -9.5 (9.2) | -10.1 (8.6)

LIMITATIONS AND CAVEATS:
Safety has been reported in the literature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes